CLINICAL TRIAL: NCT00387075
Title: Parkinson Associated Risk Factor Study (PARS): Evaluating Potential Screening Tools for Parkinson Disease
Brief Title: A Study Evaluating Potential Screening Tools for Detecting Parkinson Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Molecular NeuroImaging (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: PARS
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; SPECT imaging
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and Investigators were not provided results of the University of Pennsylvania Smell Identification Test (UPSIT).
Oversight: Data Monitoring Committee: No

ARMS (1):
- [123I]β-CIT and SPECT imaging (Experimental): To Assess [123I]β-CIT and SPECT imaging
  Interventions: Procedure: [123I]β-CIT and SPECT imaging; Drug: [123I]β-CIT

INTERVENTIONS:
Procedure: [123I]β-CIT and SPECT imaging — This study is designed as a prospective cohort study to test the strategy of combining two biomarkers of parkinsonism, olfaction and brain imaging with a radioactively labeled drug, [123I]β-CIT , in a population of first-degree relatives of PD patients as a tool to establish an 'at risk' Parkinson disease cohort without motor symptoms of PD.
Drug: [123I]β-CIT — SPECT imaging uses the single photon emissions from radioactive compounds that are (most commonly) injected into a patient and are metabolized by specific organs or body systems. SPECT imaging is performed by using a gamma camera to acquire multiple 2-D images (also called projections),

SUMMARY:
This study is designed as a prospective cohort study to test the strategy of combining two biomarkers of parkinsonism, olfaction and brain imaging with a radioactively labeled drug, [123I]β-CIT , in a population of first-degree relatives of PD patients as a tool to establish an 'at risk' Parkinson disease cohort without motor symptoms of PD. First-degree relatives of PD will be recruited through PD research sites and national foundations to participate in this study. In addition, first degree relatives of PD patients will be recruited directly through advertising.

DETAILED DESCRIPTION:
First-degree relatives that agree to participate (n=3,000) will be asked to complete a 40-item olfactory identification test provided by mail. 300 subjects (225 with decreased odor identification and 75 with normal olfaction) will be invited to undergo DAT imaging at the Institute for Neurodegenerative Disorders in New Haven, CT. There will also be additional clinical follow-up at participant's clinical (local) site. The primary outcome measure for the study will be the mean striatal uptake of [123I]B-CIT in first-degree relatives with a loss of odor identification, which will be compared to an established healthy control database (age 40-70; n=50). 300 relatives will be followed longitudinally with clinical evaluations and a second imaging study completed after two years. Comparing the first and second scans in this subset of subjects will allow us to evaluate the rate of progressive loss in dopamine transporter density during this pre-symptomatic period.

ELIGIBILITY:
At Risk - Inclusion Criteria:

* subject must have a first-degree relative with PD, based on their report
* subject must not carry a diagnosis of PD or other neurodegenerative disorder.
* subject must be either at least 50 yrs old or within 10 yrs of the age of onset of their affected relative
* Subject must have no other known reason for abnormal olfaction (e.g. nasal trauma, sinus infection, sinus surgery)
* Subject must not be pregnant if participating in the imaging portion of this study

Non-First Degree Relative - Inclusion Criteria:

* Subject must not carry a diagnosis of PD or other neurodegenerative disorders
* Subject must have no other known reason for abnormal olfaction (e.g. nasal trauma, sinus infection, sinus surgery)
* Subject must not be pregnant or be an actively nursing mother if participating in the imaging portion of this study.

Exclusion Criteria:

* diagnosis of PD or other neurodegenerative disorder
* other known reason for abnormal olfaction (e.g. nasal trauma, sinus infection, sinus surgery)
* pregnancy, if participating in the imaging portion of this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2006-11; Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
the mean striatal uptake of [123I]B-CIT in first-degree relatives with a loss of odor identification, compared to an established healthy control database (age 40-70; n=50) | 1 year

SECONDARY OUTCOMES:
Estimate the frequency of olfactory loss of first-degree relatives of PD patients | 1 year
Compare striatal DAT imaging in first-degree relatives of PD patients without signs or symptoms of PD with olfactory loss to age matched healthy controls | 1 year
Determine if a reduction in DAT density using [123I]B-CIT and SPECT imaging in first-degree relatives of PD patients without signs or symptoms of PD at baseline predicts the onset of clinical PD at 2-year follow-up | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, MD, PhD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Morrish PK, Rakshi JS, Bailey DL, Sawle GV, Brooks DJ. Measuring the rate of progression and estimating the preclinical period of Parkinson's disease with [18F]dopa PET. J Neurol Neurosurg Psychiatry. 1998 Mar;64(3):314-9. doi: 10.1136/jnnp.64.3.314. PMID 9527140
- [Background] Fearnley JM, Lees AJ. Ageing and Parkinson's disease: substantia nigra regional selectivity. Brain. 1991 Oct;114 ( Pt 5):2283-301. doi: 10.1093/brain/114.5.2283. PMID 1933245
- [Background] DeKosky ST, Marek K. Looking backward to move forward: early detection of neurodegenerative disorders. Science. 2003 Oct 31;302(5646):830-4. doi: 10.1126/science.1090349. PMID 14593169
- [Background] Braak H, Del Tredici K, Rub U, de Vos RA, Jansen Steur EN, Braak E. Staging of brain pathology related to sporadic Parkinson's disease. Neurobiol Aging. 2003 Mar-Apr;24(2):197-211. doi: 10.1016/s0197-4580(02)00065-9. PMID 12498954
- [Background] Lang AE, Obeso JA. Challenges in Parkinson's disease: restoration of the nigrostriatal dopamine system is not enough. Lancet Neurol. 2004 May;3(5):309-16. doi: 10.1016/S1474-4422(04)00740-9. PMID 15099546
- [Derived] Brumm MC, Pierz KA, Lafontant DE, Caspell-Garcia C, Coffey CS, Siderowf A, Marek K. Updated Percentiles for the University of Pennsylvania Smell Identification Test in Adults 50 Years of Age and Older. Neurology. 2023 Apr 18;100(16):e1691-e1701. doi: 10.1212/WNL.0000000000207077. Epub 2023 Feb 27. PMID 36849448